CLINICAL TRIAL: NCT06495411
Title: "The Effect of Pranayama and Deep Breathing Exercises on Shoulder Pain and Sleep Quality After Laparoscopic Cholecystectomy"
Brief Title: Pranayama and Deep Breathing Exercises Sleep Quality After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Kurt, graduate student, Ataturk University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: Ekurt
Record Dates: First submitted 2024-06-10; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: pranayama, shoulder pain, sleep quality
MeSH Terms: conditions — Shoulder Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pranayama- (Experimental): Patients will perform breathing exercises every two hours from the 4th hour after surgery until discharge. Then, their pain will be evaluated with the Visual analog scale before and after exercise at the 6th hour, 12th hour, 24th hour and at discharge.
  Interventions: Other: pranayama-
- deep breathing - (Experimental): Patients will perform breathing exercises every two hours from the 4th hour after surgery until discharge. Then, their pain will be evaluated with the Visual analog scale before and after exercise at the 6th hour, 12th hour, 24th hour and at discharge.
  Interventions: Other: deep breathing-
- control (Experimental): Patients will not undergo any postoperative intervention. Then, their pain will be evaluated with the Visual analog scale at the 6th hour, 12th hour, 24th hour and at discharge.
  Interventions: Other: control

INTERVENTIONS:
Other: pranayama- — Pain of patients will be evaluated with the Visual analog scale at the 6th hour, 12th hour, 24th hour and at discharge.
  Other Names: PRANAYAMA
  Arms: pranayama-
Other: deep breathing- — Pain of patients will be evaluated with the Visual analog scale at the 6th hour, 12th hour, 24th hour and at discharge.
  Arms: deep breathing -
Other: control — Pain of patients will be evaluated with the Visual analog scale at the 6th hour, 12th hour, 24th hour and at discharge.
  Arms: control

SUMMARY:
This study explores the impact of pranayama and deep breathing exercises on alleviating shoulder pain and improving sleep quality following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The data were collected by the researcher by face-to-face interview method at SBU Van Training and Research Hospital General Surgery Clinics. Necessary information was given to healthcare professionals in the clinics where the research would be conducted, and the lists of patients who would undergo surgery were followed. Data collection started in the preoperative period, and the data collection phase ended when the patient was discharged after the surgery.

To collect pranayama, deep breathing and control group data, the researcher identified patients who were scheduled to undergo laparoscopic cholecystectomy surgery in general surgery services on a daily basis and met the sampling criteria. In the hospital where the research was conducted, laparoscopic cholecystectomy surgeries were performed excluding emergency surgeries.

It is performed electively and patient education is provided on the day of surgery. Patients are taken into surgery according to the surgery list determined the day before.

It was determined by randomization whether the patients participating in the study would be in the control or experimental groups. Patients were included in the study according to randomization order. Patients coming for surgery were randomly assigned to a pranayama group, a deep breathing group, and a control group.

This randomization technique was continued until the sample number in the research groups was reached, and the study was terminated when 22 patients were included in the pranayama group, 22 in the deep breathing group and 22 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain after elective laparoscopic cholecystectomy surgery patients,
* No hearing-speech problems that would hinder communication,
* No cognitive-mental problems,
* Not having any psychiatric disease,
* No sleep disorder
* Patients who have not previously attended courses on breathing exercises and yoga,
* All volunteers who agreed to participate in the study were included in the study.

Exclusion Criteria:

* Admitted to the intensive care unit in the early postoperative period,
* Extra surgical intervention (hernia repair, etc.),
* During laparoscopic cholecystectomy, patients undergoing open cholecystectomy patients were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain after laparoscopic cholecystectomy with visual analogue scale in deep breathing group, pranayama group and control groups. | Pain was evaluated before surgery. After surgery, pain was evaluated before and after exercise, at the 6th hour, 12th hour, 24th hour and at discharge.
  On the visual analogue scale, 0 points mean no pain, and 10 points mean unbearable pain.

SECONDARY OUTCOMES:
Evaluation of sleep of patients after laparoscopic cholecystectomy with the Richard Campbell Sleep Scale | The sleep quality of the patients was measured before the surgery and in the morning of the second day of the surgery.
  Sleep is evaluated on a chart between 0 and 100. A score between "0-25" from the scale indicates very poor sleep, and a score between "76-100" indicates very good sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Kurt E, Yayla A. The Effects of Pranayama and Deep Breathing Exercises on Pain and Sleep Quality After Laparoscopic Cholecystectomy. Nurs Health Sci. 2025 Mar;27(1):e70041. doi: 10.1111/nhs.70041. PMID 39870367